CLINICAL TRIAL: NCT06635941
Title: A Predictive Model Identifies Patients Likely To Be Painful During Sedation-free Colonoscopy.
Brief Title: Predictive Model Identifies Painful Sedation-free Colonoscopy
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-110A-01
Record Dates: First submitted 2024-09-22; First posted 2024-10-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Pain; Non-sedated; Colonoscopy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer is one of the most common cancers globally and a leading cause of cancer-related death. Colonoscopy is the standard screening method for colorectal cancer, significantly reducing mortality rates. However, the pain experienced during the procedure is one of the main reasons people avoid getting a colonoscopy. If operators can identify patients who are more likely to feel pain before the procedure, operators can take steps to reduce their discomfort. Previous research has developed a model to predict discomfort during colonoscopy, but this model have some limitations in clinical use. Therefore, investigators plan to develop a new model that also predicts the likelihood of painful colonoscopies.

This study aims to identify factors related to pain in non-sedated colonoscopy and create a more accurate prediction model to help reduce pain during the procedure.

A total of 679 patients will be divided into two groups randomly for training and validation. Participants meet the inclusion criteria for this study, and investigators will ask participants to participate voluntarily. If participants agree, investigators will collect some of participants basic information and medical history, and assess participants' pain during the procedure.

Participants will only need to follow the doctors' instructions, complete bowel investigators' preparation, and undergo the colonoscopy as usual. The data collection will not interfere with participants' regular care

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing non-sedated colonoscopy at Ningbo University Affiliated Hospital from September 2024 to September 2025.
2. Age: Patients aged 18 to 75 years.
3. Voluntary participation: Patients who voluntarily agree to participate in the study and have signed the informed consent form.

Exclusion Criteria:

1. Patients under 18 years old.
2. Patients who are unwilling or unable to provide informed consent.
3. Patients with malignant diseases, severe chronic heart or lung diseases, or those who have received treatment or radiation therapy for coronary artery or cerebrovascular events requiring hospitalization in the past 3 months.
4. Patients with a history of colorectal resection or those with an incomplete colon.
5. Patients who do not require reaching the ileocecal valve.
6. Patients who have not completed bowel preparation or who have only used enemas for bowel cleaning.
7. Patients with severe bowel obstruction or bowel perforation.
8. Pregnant or breastfeeding women. -

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: the people who is about to have a sedation-free colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-09-21 (Actual); Study Completion 2025-09-21 (Actual)

PRIMARY OUTCOMES:
colonoscopy-related pain | during the intubation procedure of sedated-free colonoscopy
  The primary outcome is the the pain during the procedure of sedated-free colonoscopy according to a 4-point verbal rating scale (VRS-4), which is a four-category lanuage scale that classifies pain as no(0), slight(1), moderate(2), and se vere(3).

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Ningbo University, Ningbo, Ningbo, Zhejiang, China